CLINICAL TRIAL: NCT03169816
Title: Lorcaserin in Combination With XR-Naltrexone for Relapse Prevention in Opioid Use Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7501
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorcaserin (Experimental): 10 mg capsule taken twice daily of lorcaserin
  Interventions: Drug: Lorcaserin
- Placebo (Placebo Comparator): a placebo comparator capsule taken twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin 10mg, twice daily
  Arms: Lorcaserin
Drug: Placebo — Matched placebo for lorcaserin condition dosed twice daily
  Arms: Placebo

SUMMARY:
This study proposes to recruit patients with Opioid Use Disorder (OUD) seeking treatment into our program of outpatient detoxification and naltrexone induction followed by a relapse-prevention treatment with Extended release-naltrexone (XR-NTX) . Eligible participants will be randomly assigned to adjunctive treatment with lorcaserin (N = 40), or placebo (N = 20) with weekly therapy.

DETAILED DESCRIPTION:
The study proposes to recruit patients with Opioid Use Disorder (OUD) seeking treatment into our program of outpatient detoxification and naltrexone induction followed by a relapse-prevention treatment with Extended release-naltrexone (XR-NTX) . Eligible participants will be randomly assigned to adjunctive treatment with lorcaserin (N = 40), or placebo (N = 20) with weekly therapy. Lorcaserin or placebo 10 mg bid will be started on Day 1 of the study to address acute withdrawal, then maintained over the next 5 weeks, and stopped after the second XR-naltrexone is administered. Patients will be seen twice weekly for monitoring and offered two injections of naltrexone; at the end of oral naltrexone induction (end of week 1) and four weeks later (week 5). The primary outcome measures will be the proportion of patients successfully inducted onto XR-naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* 1. Individuals between the ages of 18-60

  2. Meets DSM-5 criteria of current opioid use disorder present for at least six months, supported by a positive urine for opioids

  3. Seeking treatment for opioid use disorder

  4. Capable of giving informed consent and complying with study procedures

  5. Not underweight; defined as BMI≥18.5

Exclusion Criteria:

1. Lifetime history of DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
2. Current DSM-5 criteria for any other psychiatric disorder that in the investigator's judgment is unstable, would be disrupted by the study medication, or is likely to require pharmacotherapy or psychotherapy during the study period. Concurrent treatment with other psychotropic medication is exclusionary.
3. Individuals who meet DSM-5 criteria for any substance use disorders - severe, other than opioid and nicotine use disorder. Physiological dependence on alcohol or sedative-hypnotics is exclusionary.
4. A recent history of binge-use of alcohol or sedative-hypnotics (using large amounts in a short time to severe intoxication or blackouts).
5. Pregnancy, lactation, or failure to use adequate contraceptive method in female patients who are currently engaging in sexual activity with men.
6. Unstable medical conditions, such as AIDS, cancer, uncontrolled hypertension (blood pressure > 140/90), uncontrolled diabetes, pulmonary hypertension or heart disease.
7. Legally mandated to participate in a substance use disorder treatment program.
8. Current or recent history of significant violent or suicidal behavior, risk for suicide or homicide
9. Currently meets DSM-5 diagnosis for an eating disorder with low body weight (BMI <20)
10. History of accidental opioid overdose in the last three years or any other significant history of overdose following detoxification within past 10 years defined as an episode of opioid-induced unconsciousness, whether or not medical treatment was sought or received.
11. Elevated liver function tests (AST and ALT > 3 times the upper limit of normal) or impaired renal function (GFR<60 ml/min)
12. Known history of allergy, intolerance, or hypersensitivity to lorcaserin, naltrexone or any other study medications
13. Concurrent use of migraine medications containing ergotamine (Cafergot, Ergomar) or dihydroergotamine (Migranal), 5HT2B receptor agonists like cabergoline, or medications metabolized by CYP2D6 (thioridazine, tamoxifen, metoprolol, aripiprazole, codeine)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, MD, Principal Investigator — NYSPI
Locations (1):
- Substance Treatment and Research Service (STARS), Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 patients were enrolled in the trial but of these 49 patients were randomized to one of the treatment arms.
Period: Overall Study
Arm/Group | Lorcaserin | Placebo
Started | 33 | 16
Completed | 6 | 3
Not Completed | 27 | 13

BASELINE CHARACTERISTICS:
Population: Baseline analysis for the 49 randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorcaserin | Placebo | Total
Number analyzed (Participants) | 33 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (9.9) | 39.5 (12.6) | 37.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 25 | 13 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 26 | 14 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 22 | 10 | 32
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Successfully Inducted to Receive Naltrexone Injection
Description: proportion of individuals who were successfully inducted and received the first XR-naltrexone injection
Time Frame: Study week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 33 | 16
Participants | 12 | 7

ADVERSE EVENTS:
Time Frame: During the 8 weeks of the trial or length of participant's participation.
Arm/Group | Lorcaserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/33 | 0/16
Other Adverse Events (participants affected / at risk) | 14/33 | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin (N=33) | Placebo (N=16)
Inpatient rehabilitation (General disorders) | 2 (2) | 0 (0) — Two participants voluntarily entered inpatient rehabilitation programs prior to completing the trial.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin (N=33) | Placebo (N=16)
insomnia (General disorders) | 3 (3) | 3 (3)
GI Upset (Gastrointestinal disorders) | 4 (4) | 1 (1)
Anorexia (General disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hot flashes (Gastrointestinal disorders) | 2 (2) | 0 (0)
Precipitated Withdrawal (General disorders) | 1 (1) | 1 (1)
Bachache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blackout (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fainting (General disorders) | 1 (1) | 0 (0)
Gout (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Head Sensation (General disorders) | 1 (1) | 0 (0)
Irritable (General disorders) | 1 (1) | 0 (0)
Leg Cramps (General disorders) | 1 (1) | 0 (0)
Loss of Libido (General disorders) | 1 (1) | 0 (0)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sexual Dysfunction (General disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
GI Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03169816/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03169816/SAP_001.pdf